CLINICAL TRIAL: NCT06293937
Title: Impact of Front-of-package Labels on Weight Bias Among Latine and Limited English Proficiency Populations
Brief Title: Impact of Front-of-package Labels on Weight Bias Among Latines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0300b
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-08

CONDITIONS: Weight Prejudice
MeSH Terms: conditions — Weight Prejudice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Numerical label (Experimental)
  Interventions: Behavioral: Numerical label
- Interpretive text-only label (Experimental)
  Interventions: Behavioral: Interpretive text-only label
- Interpretive magnifying glass icon label (Experimental)
  Interventions: Behavioral: Interpretive magnifying glass icon label
- Separated interpretive magnifying glass icon label (Experimental)
  Interventions: Behavioral: Separated interpretive magnifying glass icon label

INTERVENTIONS:
Behavioral: Numerical label — Labels that list the amount and percent of daily value of added sugar, sodium, or saturated fat, modeled after Guideline Daily Amounts labels.
  Arms: Numerical label
Behavioral: Interpretive text-only label — Interpretive text-only labels that state when a product contains high amounts of added sugar, sodium, or saturated fat.
  Arms: Interpretive text-only label
Behavioral: Interpretive magnifying glass icon label — Interpretive labels that state when a product contains high amounts of added sugar, sodium, or saturated fat, containing a magnifying glass icon.
  Arms: Interpretive magnifying glass icon label
Behavioral: Separated interpretive magnifying glass icon label — Interpretive labels that state when a product contains high amounts of added sugar, sodium, or saturated fat, containing a magnifying glass icon. Each nutrient will be on a separate label.
  Arms: Separated interpretive magnifying glass icon label

SUMMARY:
The goal of this experiment is to examine the effects on explicit weight bias of a selection task using 4 different types of front-of-package food labels to select healthy or unhealthy foods among a sample of Latine and low English proficiency adults. The main questions this experiment aims to answer are:

* Does the use of different front-of-package label designs in a selection task lead to different effects on explicit weight bias among Latine and low English proficiency consumers?
* Does the use of different front-of-package label designs in a selection task lead to different effects on attribution of personal responsibility for body weight among Latine and low English proficiency consumers?

Participants will be randomly assigned to 1 of 4 types of front-of-package label designs. They will view 3 sets of products (frozen meals, frozen pizzas, and frozen desserts), shown in random order. For each product set, participants will view 3 products shown in random arrangement, each with participants' randomly assigned label shown on the front of package. After viewing all 3 product types, participants will answer questions about explicit weight bias and attribution of responsibility for body weight. Researchers will compare results across label designs.

DETAILED DESCRIPTION:
This study aims to determine if the use of different front-of-package label types in a selection task leads to different effects on explicit weight bias and attribution of responsibility for body weight among Latine and low English proficiency (LEP) consumers. A Latine-focused panel company will recruit 4,000 US Latine adults of parental age (18-55 years), approximately 50% of whom will have low English proficiency (LEP). In a between-subjects experiment, researchers will randomize participants to 1 of 4 types of front-of-package labels: a numerical label, an interpretive text-only label, an interpretive label with a magnifying glass icon, or separated interpretive labels with a magnifying glass icon. Participants will first perform a selection task for a parent study in which they will view their assigned label on 3 sets of products (with 3 products per set) and select the product they believe is most and least healthy and the product they most want to purchase. After this selection task, participants will answer questions measuring this study's outcomes: explicit weight bias (primary outcome) and attribution of personal responsibility of body weight (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Identifying as Latine or Hispanic
* Ages 18-55 years old
* Residing in the United States

Exclusion Criteria:

* Not identifying as Latine or Hispanic
* Less than 18 or greater than 55 years old
* Not residing in the United States

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3306 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Explicit weight bias, mean score | Immediately after exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Explicit weight bias will be measured by survey through a six-item scale. Items will present participants with adjective pairs and ask that they select the box closest to the adjective that they feel best describes their feelings and beliefs about people with obesity: (1) lazy - hard-working, (2) no will power - has will power, (3) good self - control - poor self-control, (4) active - inactive, (5) dislikes food - likes food, (6) undereats - overeats. Response options, which will be presented as 5 boxes between adjectives, will be coded in a categorical 1-5 range where higher scores represent higher endorsement of a stereotype that contributes to weight bias. Each participant's responses to each item will then be averaged across the 7 items to obtain their final score on the outcome in a 1-5 range, where higher scores represent higher explicit weight bias.

SECONDARY OUTCOMES:
Attribution of personal responsibility for body weight, mean score | Immediately after exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Attribution of personal responsibility for body weight will be measured by survey through a two-item scale. Items will ask participants how much they agree with two statements: (1) People with obesity are responsible for their weight; (2) People with obesity are to blame for their weight. Response options will be on a 5-point scale from strongly disagree to strongly agree, with higher scores representing higher agreement. Each participant's responses to each item will be averaged to obtain their final score on the outcome in a 1-5 range, where higher scores represent higher attribution of personal responsibility for body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Aline D'Angelo Campos, MPP, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill's Gillings School of Global Public Health, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan will be shared prior to data collection. After data collection and analysis, a de-identified version of individual participant data and the analytic code will be shared through the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Study Protocol and SAP will be available by mid-March 2024 (prior to data collection). IPD and analytic code will become available after data collection and analysis.
Access Criteria: Open access.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT06293937/Prot_SAP_000.pdf